CLINICAL TRIAL: NCT01360762
Title: Secondary Prophylaxis of Visceral Leishmaniasis Relapses in HIV Co-infected Patients Using Pentamidine as a Prophylactic Agent: a Prospective Cohort Study
Brief Title: Prophylaxis of Visceral Leishmaniasis Relapses in HIV Co-infected Patients With Pentamidine: a Cohort Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Addis Ababa University (Other); University of Gondar (Other); Tigray Regional Health Bureau, Tigray Region (Unknown); Amhara Regional Health Bureau, Amhara Region (Unknown); Medecins Sans Frontieres, Netherlands (Other); Leishmania East Africa Platform (LEAP) (Unknown); Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ITMC0109
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Visceral Leishmaniosis; HIV-infection/Aids
Keywords: Secondary prophylaxis; Visceral leishmaniasis; Relapses; HIV co-infection; Pentamidine; Ethiopia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Leishmaniasis, Visceral; Recurrence | interventions — Pentamidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pentamidine Secondary Prophylaxis (PSP) (Experimental): Patients with co-infection of human immunodeficiency virus (HIV)and visceral leishmaniosis (VL), having being treated for VL, are allocated to pentamidine secondary prophylaxis, to prevent VL relapses. The treatment period is of 12 months, plus an "extended treatment period" of 0 to 6 months depending on the immunosuppression status, plus 12 months follow-up after the extended treatment period.
  Interventions: Drug: Pentamidine

INTERVENTIONS:
Drug: Pentamidine — Pentamidine isethionate 300 mg for one vial for intramuscular or intravenous route(1 mg of pentamidine isethionate is equivalent to 0.57 mg of pentamidine base)
  Other Names: PENTACARINAT 300 mg, by Sanofi-Aventis

SUMMARY:
Visceral leishmaniosis (VL) is widely reported in Ethiopia, with about 30% of cases being associated with human immunodeficiency virus (HIV). In absence of antiretroviral treatment (ART), poor prognosis, high mortality and high relapse rates are characteristic of Ethiopian VL patients with HIV co-infection. Conversely, co-infection can be successfully managed via a combination of effective treatment of the initial episode, timely ART and prevention of relapses.

Actually, until cellular immunity returns with ART, the patient is at risk of VL relapses, which can result in death, severe illness, reduced ART efficacy, drug-resistance and possibly transmission of drug-resistant Leishmania donovani. Patients most vulnerable to relapses are those with high levels of immunosuppression, with previous VL episodes, or with opportunistic infections (OIs). The most important factor to prevent relapses seems to be the clearance of visible parasites.

Limited studies in Europe show that HIV co-infected patients may benefit from secondary prevention with antimonials (part of mainstay treatment for VL in Ethiopia) and pentamidine (PM), not used for VL treatment in Africa. Such maintenance treatment has not been studied in African VL, but the poor outcomes without secondary prevention highlight a need of better care to patients at risk of relapse.

This prospective cohort study aims at documenting the patient's outcomes of secondary prophylaxis with PM in VL-HIV co-infection, in terms of time to relapse or death, safety and feasibility, before it can be considered for general use in Ethiopia. A placebo group is not included, due to the clear advantages of the intervention to the patient population.

DETAILED DESCRIPTION:
Visceral leishmaniosis (VL) in Ethiopia has been reported in different parts of the country, with approximately 30% of cases being associated with human immunodeficiency virus (HIV). The ruralisation of HIV epidemic in VL endemic areas will hamper efforts to control VL. Clinical experience in Ethiopia has shown that anti-leishmanial treatment in the absence of anti-retroviral therapy (ART) does not result in favourable outcomes: poor prognosis, high mortality and relapse rates are characteristic of Ethiopian VL patients with HIV co-infection. The effective management of the initial VL episode, timely ART, and prevention of relapses should be the cornerstones of effective management of HIV/VL co-infection.

However, parasitological cure of VL in HIV co-infected patients cannot easily be established, and until cellular immunity returns with ART, the patient is at risk of relapses of VL, which can result in death, severe illness, negative effect on ART efficacy leading to other opportunistic infections (OIs), emergence of drug-resistant parasites, and possibly to transmission of drug-resistant Leishmania donovani. Patients most vulnerable to relapses are 1) those with high levels of immunosuppression, 2) patients with previous VL episodes, and 3) patients with OIs.

ART reduces the risk of VL relapse/recurrence by ~50%, while the type of anti-leishmanial primary treatment has little effect on relapses; the most important factor seems to be clearance of visible parasites (if residual parasites are seen at the end of treatment, the relapse rate is 100%).

Limited studies in Europe show that HIV co-infected patients may benefit from secondary prevention, by significantly prolonging the relapse-free period. The drugs studied for secondary prophylaxis in Europe have been meglumine antimoniate and AmBisome, which are part of mainstay treatment for VL in Ethiopia, and pentamidine (PM), which is not used for VL treatment in Africa. The effect of such maintenance treatment has not been studied in African VL, but the poor outcomes without secondary prevention highlight a clear need to offer better care to patients at high risk of relapse.

Indeed, secondary prophylaxis is generally recommended in Europe and the United States (see the 2009 Center for Disease Control guidelines). PM 4 mg/kg intravenous (IV) every 3-4 weeks has been proposed as secondary prophylaxis, and it is already used in countries like United Kingdom and Spain.

Consequently, this prospective cohort study aims at documenting the patient's outcomes of secondary prophylaxis with PM in VL-HIV co-infection, in terms of time to relapse or death, safety and feasibility, before it can be considered for more general use in Ethiopia. A placebo group is not included, due to the clear advantages of the intervention to the patient population targeted herewith. Furthermore as other available VL treatments are used as main line treatments, they cannot be considered as alternative comparators, given the potential risk of rapid emergence of drug resistance and subsequent spread in areas of anthroponotic VL.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Visceral Leishmaniosis (VL) during the recruitment period that are EITHER treated for VL relapse and have a documented negative test of cure (TOC), OR are treated for primary VL and have a documented CD4 <200 or WHO stage 4 disease during the recruitment period and have a documented negative TOC
* Patients treated for VL in the past with documented CD4 <200 or WHO stage 4 disease during the recruitment period AND documented negative TOC after the latest VL treatment and currently asymptomatic OR currently negative diagnostic test (microscopy)
* Patients agreeing to start or continue antiretroviral treatment (first or second line)
* Patients willing to provide written informed consent

Exclusion Criteria:

* Patients with known hypersensitivity to pentamidine
* Patients with known renal failure
* Patients with diabetes mellitus (type I or II)
* Patients unlikely to attend follow-up visits/comply with study requirements
* Pregnant and lactating women
* Any other condition that could increase the risk of toxicity of pentamidine to such an extent outweighing the expected benefit (eg severe cardiac dysfunction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ermias Diro, MD, Study Director — University of Gondar, Ethiopia; Johan Van Griensven, MD, PhD, Study Director — ITM
Locations (3):
- Ethiopia (3):
  - Abdurafi Health Center/Médecins Sans Frontières, Abdurafi, Amhara
  - Kahsay Abera Hospital, Humera, Tigray
  - Leismania Research and Treatment Centre, University of Gondar Hospital, Gonder

REFERENCES:
- [Derived] Diro E, Ritmeijer K, Boelaert M, Alves F, Mohammed R, Abongomera C, Ravinetto R, De Crop M, Fikre H, Adera C, van Loen H, Tsoumanis A, Adriaensen W, Hailu A, Griensven JV. Long-term Clinical Outcomes in Visceral Leishmaniasis/Human Immunodeficiency Virus-Coinfected Patients During and After Pentamidine Secondary Prophylaxis in Ethiopia: A Single-Arm Clinical Trial. Clin Infect Dis. 2018 Jan 18;66(3):444-451. doi: 10.1093/cid/cix807. PMID 29020217

RESULTS

PARTICIPANT FLOW:
Groups:
- Pentamidine Secondary Prophylaxis (PSP): Patients with co-infection of human immunodeficiency virus (HIV) and visceral leishmaniosis (VL), having being treated for VL.
Period: Main Study Period (12-month Treatment)
Arm/Group | Pentamidine Secondary Prophylaxis (PSP)
Started | 74
Completed | 45
Not Completed | 29
Not completed — Lost to Follow-up | 7
Not completed — Death | 5
Not completed — Discontinuation of study drug for safety | 1
Not completed — Patient relapsed | 15
Not completed — Discontinuation | 1
Period: Whole Study Period
Arm/Group | Pentamidine Secondary Prophylaxis (PSP)
Started (Treatment period and extended treatment period and follow-up period) | 74
Completed | 38
Not Completed | 36
Not completed — Lost to Follow-up | 10
Not completed — Death | 7
Not completed — Patient relapsed | 18
Not completed — Discontinuation of study drug for safety | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pentamidine Secondary Prophylaxis (PSP)
Number analyzed (Participants) | 74
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [28 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 71
Weight [Median (Inter-Quartile Range); unit: kg] | 50 [44.6 to 53]
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  BMI < 18.5 kg/m^2 | 56
  BMI > 18.5 kg/m^2 | 18
Functional status [Count of Participants; unit: Participants] — Population: Information for one participant is missing.
  Participants
    number analyzed (Participants) | 73
    Working | 46
    Ambulatory | 25
    Bed ridden | 2
Spleen size [Count of Participants; unit: Participants] — Population: 1 Subjects had no spleen size calculation due to ascites.
  Participants
    number analyzed (Participants) | 73
    not palpable | 30
    Palpable < 5 cm | 14
    Palpable 5 cm or > 5 cm | 29
Total liver span [Median (Inter-Quartile Range); unit: cm] | 11 [10 to 13]
Total WBC count [Median (Inter-Quartile Range); unit: cells/µL] | 3000 [2300 to 3900]
Neutrophil percent [Median (Inter-Quartile Range); unit: percentage of neutrophils] | 62.3 [48.4 to 70.6]
Lymphocyte percent [Median (Inter-Quartile Range); unit: percentage of lymphocytes] | 27.8 [21.9 to 38.5]
Haemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 9.2 [7.7 to 11.1]
Platelet count [Median (Inter-Quartile Range); unit: platelets x10^3 / µL] | 192 [136 to 274]
Current CD4 count [Median (Inter-Quartile Range); unit: cells/µL] | 127 [85 to 185]
Current CD4 count [Count of Participants; unit: Participants]
  50 or less | 7
  51-100 | 15
  101-200 | 37
  201-350 | 7
  more than 350 | 5
  Missing | 3
VL status [Count of Participants; unit: Participants] — status of visceral leishmaniasis (primary infection or relapse)
  Participants
    Primary | 31
    Relapse | 43
Number of VL episodes before inclusion [Count of Participants; unit: Participants] — Population: There were only 43 subjects out of the 74 total population that were relapse subjects. The other 31 subjects had a primary infection
  Participants
    number analyzed (Participants) | 43
    1 episode | 27
    2 episodes | 12
    3 episodes | 3
    4 episodes | 1

OUTCOME MEASURES:

1. Primary Outcome: Probability of Relapse-free Survival
Description: Probability of relapse-free survival up to one year after the start of the intervention (PSP) (at month 6 and month 12)
Time Frame: up to 1 year after the start of the intervention (PSP)
Measure: Number (95% Confidence Interval); unit: percentage probability
Arm/Group | Pentamidine Secondary Prophylaxis (PSP)
Number analyzed (Participants) | 74
percentage probability
  Probability of relapse-free survival at 6 months | 79 [67 to 87]
  Probability of relapse-free survival at 12 months | 71 [59 to 80]

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of patients with SAEs which are possibly, probably or definitely drug-related following clinician's assessment or that lead to permanent drug discontinuations during the first year of pentamidine administration
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pentamidine Secondary Prophylaxis (PSP)
Number analyzed (Participants) | 74
Participants | 3

3. Secondary Outcome: Number of Participants With Adverse Events
Description: During the first year of pentamidine administration for prophylaxis: participants with any drug-related non-serious adverse events (with drug-related defined as possibly, probably or definitely related to primary therapy following physicians assessment) as well as any serious adverse events (drug-related or not)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pentamidine Secondary Prophylaxis (PSP)
Number analyzed (Participants) | 74
Participants
  Drug-related non-serious adverse events | 30
  Any serious adverse event | 17

4. Secondary Outcome: Number of Treatment Discontinuations and Interruptions
Description: Number of treatment discontinuations and interruptions/missed doses.
Time Frame: 30 months
Measure: Number; unit: number of events
Arm/Group | Pentamidine Secondary Prophylaxis (PSP)
Number analyzed (Participants) | 74
number of events
  Permanent discontinuation | 2
  Missed more than 1 dose | 4
  Treatment interruption | 0

5. Secondary Outcome: Number of Required Additional Interventions
Description: The number of required additional clinical interventions/therapeutic procedures
Time Frame: 30 months
Measure: Number; unit: number of events
Arm/Group | Pentamidine Secondary Prophylaxis (PSP)
Number analyzed (Participants) | 74
number of events
  Additional IV fluid during PM administration | 10
  Prolonged hospital observation | 2
  additional medication during PM infusion | 2
  Additional IV or oral glucose | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the whole study period of 30 months (primary study period (12 months), extended study period (6 months) and 12 months follow-up period).
Arm/Group | Pentamidine Secondary Prophylaxis (PSP)
All-Cause Mortality (participants affected / at risk) | 7/74
Serious Adverse Events (participants affected / at risk) | 33/74
Other Adverse Events (participants affected / at risk) | 71/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pentamidine Secondary Prophylaxis (PSP) (N=74)
Diarrhoea (Gastrointestinal disorders) | 1
Upper gastro-intestinal haemorrhage (Gastrointestinal disorders) | 1
Disseminated tuberculosis (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Bacterial Lymphadenitis (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 16
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Hypovolemic shock (Blood and lymphatic system disorders) | 2
Uveitis (Eye disorders) | 1
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Giardiasis (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Tuberculosis of central nervous system (Infections and infestations) | 1
Typhoid fever (Infections and infestations) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Demyelinating polyneuropathy (Nervous system disorders) | 1
Acute renal failure (Renal and urinary disorders) | 1
Visceral Leishmaniasis (Infections and infestations) | 20
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pentamidine Secondary Prophylaxis (PSP) (N=74)
Anaemia (Blood and lymphatic system disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 11
Gastritis (Gastrointestinal disorders) | 9
Hemorrhoids (Gastrointestinal disorders) | 4
Peptic ulcer (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 5
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1
Cataract (Eye disorders) | 1
Allergic conjunctivitis (Eye disorders) | 1
Eye allergy (Eye disorders) | 2
Eye degenerative disorder (Eye disorders) | 1
Iridocyclitis (Eye disorders) | 3
Night blindness (Eye disorders) | 2
Ocular hyperaemia (Eye disorders) | 2
Refraction disorder (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Abdominal distention (Gastrointestinal disorders) | 1
Upper abdominal pain (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Haemorrhagic diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Pancreatitis (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 4
Upper gastrointestinal haemorrhagues (Gastrointestinal disorders) | 2
Application site hypersensitivity (General disorders) | 2
Asthenia (General disorders) | 1
Chest pain (General disorders) | 10
Chills (General disorders) | 1
Injection site hypersensitivity (General disorders) | 2
Local swelling (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 10
Cholecystitis acute (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Abscess limb (Infections and infestations) | 1
Abscess neck (Infections and infestations) | 1
Acarodermatitis (Infections and infestations) | 1
Acute tonsillitis (Infections and infestations) | 1
Amoebiasis (Infections and infestations) | 6
Amoebic dysentery (Infections and infestations) | 2
Anal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Ascariasis (Infections and infestations) | 2
Atypical pneumonia (Infections and infestations) | 7
Body tinea (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 4
Bronchopneumonia (Infections and infestations) | 1
Carbuncle (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 4
Cerebral toxoplasmosis (Infections and infestations) | 2
Cestode infection (Infections and infestations) | 4
Chlamydial infection (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Disseminated tuberculosis (Infections and infestations) | 1
Dysentery (Infections and infestations) | 9
Eye infection (Infections and infestations) | 2
Bacterial eye infection (Infections and infestations) | 7
Folliculitis (Infections and infestations) | 2
Fungal skin infection (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 16
Giardiasis (Infections and infestations) | 14
Helminthic infection (Infections and infestations) | 7
Viral hepatitis (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 6
Hookworm infection (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Impetigo (Infections and infestations) | 3
Influenza (Infections and infestations) | 1
Intertrigo candida (Infections and infestations) | 2
Isopsoriasis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Lymph node tuberculosis (Infections and infestations) | 1
Bacterial lymphadenitis (Infections and infestations) | 1
Malaria (Infections and infestations) | 19
Meningitis (Infections and infestations) | 1
Nasopharingitis (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 3
Oral herpes (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Acute otitis media (Infections and infestations) | 1
Periorbital cellulitis (Infections and infestations) | 1
Bacterial peritonitis (Infections and infestations) | 1
Plasmodium falciparum infection (Infections and infestations) | 3
Plasmodium vivax infection (Infections and infestations) | 8
Pneumonia (Infections and infestations) | 32
Pulmonary tuberculosis (Infections and infestations) | 1
Pulpitis dental (Infections and infestations) | 1
Pyomyositis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Strongyloidiasis (Infections and infestations) | 3
Subcutaneous abscess (Infections and infestations) | 1
Syphilis (Infections and infestations) | 1
Taeniasis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 3
Tuberculosis of central nervous system (Infections and infestations) | 1
Typhoid fever (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 10
Visceral leishmaniasis (Infections and infestations) | 21
Wound infection (Infections and infestations) | 2
Accident at work (Injury, poisoning and procedural complications) | 1
Animal bite (Injury, poisoning and procedural complications) | 2
Chest injury (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 2
Laceration (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 2
Soft tissue injury (Injury, poisoning and procedural complications) | 4
Wound (Injury, poisoning and procedural complications) | 1
Blood albumin decreased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Creatinine renal clearance decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypovitaminosis (Metabolism and nutrition disorders) | 3
Tetany (Metabolism and nutrition disorders) | 1
Arthralgia (Metabolism and nutrition disorders) | 14
Back pain (Metabolism and nutrition disorders) | 4
Myalgia (Metabolism and nutrition disorders) | 2
Pain in extremity (Metabolism and nutrition disorders) | 3
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Demyelinating polyneuropathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 8
Migraine (Nervous system disorders) | 2
Myelopathy (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Peripheral neuropathy (Nervous system disorders) | 8
Polyneuropathy (Nervous system disorders) | 1
Post herpetic neuropathy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Somatoform disorder (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Acute renal failure (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 1
Urethral discharge (Renal and urinary disorders) | 3
Genital ulceration (Reproductive system and breast disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 1
Scrotal swelling (Reproductive system and breast disorders) | 2
Testicular swelling (Reproductive system and breast disorders) | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 16
Acne (Skin and subcutaneous tissue disorders) | 1
Cold urticaria (Skin and subcutaneous tissue disorders) | 1
Dandruff (Skin and subcutaneous tissue disorders) | 1
Allergic dermatitis (Skin and subcutaneous tissue disorders) | 3
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5
Psoriasis (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 4
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 13
Hypovolaemic shock (Vascular disorders) | 2
Shock (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes